CLINICAL TRIAL: NCT00060528
Title: A Phase I/II Pilot Study of Sequential Vaccinations With rFowlpox-PSA (L155)-TRICOM (PROSTVAC-F/TRICOM) Alone, or in Combination With rVaccinia-PSA (L155)-TRICOM (PROSTVAC-V/TRICOM), and the Role of GM-CSF, in Men With Prostate Cancer
Brief Title: Sequential Vaccinations in Prostate Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Gulley, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 030176; 03-C-0176; NCT00062153 (obsolete NCT alias)
Record Dates: First submitted 2003-05-07; First posted 2003-05-07 (Estimated); Results first posted 2012-02-23 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-09

CONDITIONS: Prostatic Neoplasms
Keywords: Immunotherapy; Cytokines; Immune Assays; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PROSTVAC; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- no GM (Experimental): No granulocyte macrophage colony stimulating factor (GM-CSF) was given
  Interventions: Drug: Recombinant Fowlpox-PSA (L155)-TRICOM (PROSTVAC-F/TRICOM)
- Rec-hGM (Experimental): Recombinant human GM-CSF (Sargramostim) was administered at 100mcg/day on days 1-4 following each vaccine. Given subcutaneously (s.c.) at site of vaccine.
  Interventions: Drug: Recombinant Vaccinia-PSA (L155)-TRICOM (PROSTVAC-V/TRICOM); Drug: Recombinant Human GM-CSF
- rF-GM (10^7pfu) (Experimental): recombinant fowlpox GM-CSF was given on day one at 10^7 in last two arms. Given subcutaneously (s.c.) at site of vaccine.
  Interventions: Drug: Recombinant Fowlpox-GM-CSF; Drug: Recombinant Fowlpox-PSA (L155)-TRICOM (PROSTVAC-F/TRICOM); Drug: Recombinant Human GM-CSF
- rF-GM (10^8) (Experimental): recombinant fowlpox GM-CSF was given on day one at 10^8 in last two arms. Given subcutaneously (s.c.) at site of vaccine.
  Interventions: Drug: Recombinant Fowlpox-GM-CSF; Drug: Recombinant Fowlpox-PSA (L155)-TRICOM (PROSTVAC-F/TRICOM); Drug: Recombinant Human GM-CSF

INTERVENTIONS:
Drug: Recombinant Fowlpox-GM-CSF
  Other Names: rF-GMCSF
  Arms: rF-GM (10^7pfu); rF-GM (10^8)
Drug: Recombinant Fowlpox-PSA (L155)-TRICOM (PROSTVAC-F/TRICOM)
  Other Names: PROSTVAC-F (fowlpox)/TRICOM
  Arms: no GM; rF-GM (10^7pfu); rF-GM (10^8)
Drug: Recombinant Vaccinia-PSA (L155)-TRICOM (PROSTVAC-V/TRICOM)
  Arms: Rec-hGM
Drug: Recombinant Human GM-CSF
  Arms: Rec-hGM; rF-GM (10^7pfu); rF-GM (10^8)

SUMMARY:
Background:

" Adenocarcinoma of the prostate is the most common cancer diagnosis in American males and follows lung cancer as the leading cause of cancer death.

" Vaccine strategies represent a novel therapeutic approach in the treatment for prostate cancer. One potential target for a prostate cancer vaccine is prostatic specific antigen (PSA), due to its restricted expression on prostate cancer and normal prostatic epithelial cells.

Objectives:

" The primary objective is to determine the impact of granulocyte-macrophage colony stimulating factor (GM-CSF) and recombinant fowlpox granulocyte-macrophage colony stimulating factor (rF-GM-CSF) on the immunologic response in patients treated with these vaccines.

" Secondary - to determine the change in prostatic specific antigen (PSA)-specific T cells in patients treated with these vaccines using enzyme linked immunosorbent spot (ELISPOT) assay analysis.

" To document any objective anti-tumor responses that may occur.

Eligibility:

" Patients must have androgen insensitive metastatic prostate cancer.

" All patients will have received and progressed on hormonal therapy.

" Must have objective evidence of metastasis or relapsing local disease. Therefore, must have a rising PSA and at least one of the following: positive bone scan, palpable disease, or positive imaging studies.

" Must have a life expectancy of more than 6 months and Eastern Cooperative Oncology Group (ECOG) status of 0 to 2.

"Patients must be human leukocyte antigen serotype within HLA-A A serotype group (HLA-A2+).

" Granulocyte count greater than or equal to 1,500/mm^3, Platelet greater than or equal to 100,000/mm^3, hemoglobin (Hgb) greater than or equal to 10Gm/dL, Lymphocyte count greater than or equal to 500/mm^3 ;Bilirubin less than 1.5mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5x upper limit of normal (ULN),Creatinine Clearance greater than or equal to 60

" No significant cardiac disease, no significant pulmonary disease, no serious inter-current medical illness.

Design:

" Cohorts three, four and five will provide safety data combining cohort two with rGM-CSF as well as two doses of rFGM-CSF respectively.

"This study will be conducted as a small, randomized pilot study to compare the immunologic effects of the above vaccine strategy alone, with recombinant granulocyte-macrophage colony stimulating factor (GM-CSF), or with either of 2 doses of fowlpox-GM-CSF.

"This study will consist of 4 randomized arms of 8 patients each, all of whom are HLA-A2+.

The maximum accrual to the trial should be 62.

DETAILED DESCRIPTION:
Background:

* Adenocarcinoma of the prostate is the most common cancer diagnosis in American males and follows lung cancer as the leading cause of cancer death.
* Vaccine strategies represent a novel therapeutic approach in the treatment for prostate cancer. One potential target for a prostate cancer vaccine is prostatic specific antigen (PSA), due to its restricted expression on prostate cancer and normal prostatic epithelial cells.

Objectives:

* The primary objective is to determine the impact of granulocyte-macrophage colony stimulating factor (GM-CSF) and recombinant fowlpox granulocyte-macrophage colony stimulating factor (rF-GM-CSF) on the immunologic response in patients treated with these vaccines.
* Secondary - to determine the change in prostatic specific antigen (PSA)-specific T cells in patients treated with these vaccines using enzyme linked immunosorbent spot (ELISPOT) assay analysis.
* To document any objective anti-tumor responses that may occur.

Eligibility:

* Patients must have androgen insensitive metastatic prostate cancer.
* All patients will have received and progressed on hormonal therapy.
* Must have objective evidence of metastasis or relapsing local disease. Therefore, must have a rising PSA and at least one of the following: positive bone scan, palpable disease, or positive imaging studies.
* Must have a life expectancy of more than 6 months and the Eastern Cooperative Oncology Group (ECOG) status of 0 to 2.
* Patients must be HLA-A2+.
* Granulocyte count greater than or equal to 1,500/mm^3, Platelet greater than or equal to 100,000/mm^3, hemoglobin (Hgb) greater than or equal to 10Gm/dL, Lymphocyte count greater than or equal to 500/mm^3; Bilirubin less than 1.5mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5x upper limit of normal (ULN),Creatinine Clearance greater than or equal to 60
* No significant cardiac disease, no significant pulmonary disease, no serious inter-current medical illness.

Design:

* Cohorts three, four and five will provide safety data combining cohort two with rGM-CSF as well as two doses of rFGM-CSF respectively.
* This study will be conducted as a small, randomized pilot study to compare the immunologic effects of the above vaccine strategy alone, with recombinant GM-CSF, or with either of 2 doses of fowlpox-GM-CSF.
* This study will consist of 4 randomized arms of 8 patients each, all of whom are HLA-A2+.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have histopathological documentation of prostate cancer confirmed in the Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI), or National Naval Medical Center (NNMC) prior to starting this study.

If no pathologic specimen is available to the NCI or NNMC, patients may enroll with a pathologist's report showing a histologic diagnosis of prostate cancer and a clinical course consistent with the disease.

Patients must have androgen insensitive metastatic prostate cancer.

Progression must be documented by at least one of the following parameters:

1. All patients must have received standard of care (hormonal) treatment before entering the trial.
2. All patients will have received and progressed on hormonal therapy for metastatic prostate carcinoma.
3. All subjects must have objective evidence of metastasis or relapsing local disease to be eligible for this Phase I trial; therefore, they must have a rising PSA and at least one of the following: positive bone scan, palpable disease, or positive imaging studies, as defined below.

i. Two consecutively rising prostatic specific antigen (PSA) levels, separated by at least 1 week, with at least one measurement that is 50% above the nadir reached after the last therapeutic maneuver (as long as the last measurement is 5 ng/ml or greater), and

ii. At least one lesion consistent with metastatic cancer on Technetium (Tc)-99 whole body scintigraphy, and/or

iii. Soft-tissue metastases as measured by appropriate modalities (i.e., imaging, palpation).

Patients must have a life expectancy of more than 6 months.

Patients must have a performance status of 0 to 2 according to the Eastern Cooperative Oncology Group (ECOG) criteria.

Patients must have recovered from any acute toxicity related to prior therapy, including surgery, and radiation (treatment must have been completed at least 4 weeks prior to being eligible for the study).

Patients who are responding to hormonal therapy are not eligible until evidence of disease progression.

Hematological eligibility parameters (within 16 days of starting therapy):

* Granulocyte count greater than or equal to 1,500/mm^3
* Platelet count greater than or equal to 100,000/mm^3
* Lymphocyte count greater than or equal to 500/mm^3
* Hemoglobin (Hgb) greater than or equal to 10 Gm/dL

Biochemical eligibility parameters (within 16 days of starting therapy):

1. A 24-hour urine collection for baseline to measure creatinine clearance (CrCl), protein and electrolytes.

   CrCl greater than 60, proteinuria less than 1000 milligrams per 24 hours, less than or equal to Grade 1 (NCI-common toxicity criteria (CTC) version 2.0) proteinuria, Grade 0 hematuria, and no abnormal sediment.

   Grade 0 creatinine.

   Patients must have serum creatinine within normal limits.

   Any abnormalities in the sediment or the presence of hematuria without a likely underlying cause should prompt the investigator to consider an evaluation by a nephrologist for evidence of underlying renal pathology. Patients may be eligible if the underlying cause of the abnormality is determined to be non-renal.
2. Hepatic function: Bilirubin less than 1.5 mg/dl,

   aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 times upper limit of normal.
3. Patients must be test negative for human immunodeficiency virus (HIV), Hepatitis B and C.

Patients must not have other active malignancies within the past 2 years (with the exception of non-melanoma skin cancers or carcinoma in situ of the bladder) or life threatening illnesses.

Patients must be willing to travel to the National Institutes of Health (NIH) for follow-up visits.

Patients must be greater than or equal to 18 years of age.

All patients who have received prior vaccination with vaccinia virus (for smallpox immunization) must not have a history of allergy or untoward reaction to the vaccine. Since vaccinia immunoglobulin (VIG) is available from the Centers for Disease Control (CDC), prior vaccinia vaccination as a safety precaution is no longer required.

Patients must understand and sign informed consent that explains the neoplastic nature of their disease, the procedures to be followed, the experimental nature of the treatment, alternative treatments, potential risks and toxicities, and the voluntary nature of participation.

Patients must not have received the following chemotherapeutic agents for cancer within 3 years of enrolling on study: docetaxel, paclitaxel, doxorubicin, cisplatinum, carboplatinum, mitoxantrone, estramustine, cyclophosphamide, irinotecan, topotecan.

Patients must not have received prior PSA vaccine therapy.

Patients will tested for human leukocyte antigen serotype within HLA-A A serotype group (HLA-A2). This test may be drawn by the patient's referring physician at the time of referral (see Appendix C, HLA-typing consent). This consent will be mailed to the patient and discussed with patient. The signed consent will be signed with a witness, then mailed to the assigned research nurse at the NIH Clinical Center. These patients must have measurable disease on computed tomography (CT), magnetic resonance imaging (MRI), or bone scan.

The effects of the study agents used in this protocol on the developing human fetus are unknown. For this reason men must agree to use adequate contraception prior to study entry and for the duration of study participation.

INCLUSION CRITERIA:

Patients must have histopathological documentation of prostate cancer confirmed in the Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI), or National Naval Medical Center (NNMC) prior to starting this study. If no pathologic specimen is available to the NCI or NNMC, patients may enroll with a pathologist's report showing a histologic diagnosis of prostate cancer and a clinical course consistent with the disease.

1. All patients will have received and progressed on hormonal therapy for metastatic prostate carcinoma.
2. All subjects must have objective evidence of metastasis or relapsing local disease to be eligible; therefore, they must have a rising PSA and at least one of the following: positive bone scan, palpable disease, or positive imaging studies, as defined below.

i. Two consecutively rising PSA levels, separated by at least 1 week, with at least one measurement that is 50% above the

nadir reached after the last therapeutic maneuver (as long as the last measurement is 5 ng/ml or greater), and

ii. At least one lesion consistent with metastatic cancer on Technetium (Tc)-99 whole body scintigraphy, and/or

iii. Soft-tissue metastases as measured by appropriate modalities (i.e., imaging, palpation).

Patients must have a life expectancy of more than 6 months.

Patients must have a performance status of 0 to 2 according to the ECOG criteria.

Patients must have recovered from any acute toxicity related to prior therapy, including surgery, and radiation (treatment must have been completed at least 4 weeks prior to being eligible for the study).

Hematological eligibility parameters (within 16 days of starting therapy):

* Granulocyte count greater than or equal to 1,500/mm^3
* Platelet count greater than or equal to 100,000/mm^3
* Lymphocyte count greater than or equal to 500/mm^3
* Hgb greater than or equal to 10 Gm/dL

Biochemical eligibility parameters (within 16 days of starting therapy):

1. A 24-hour urine collection for baseline to measure creatinine clearance (CrCl), protein and electrolytes.

   CrCl greater than 60

   proteinuria less than 1000 milligrams per 24 hours, less than or equal to Grade 1 (NCI-Common Toxicity Criteria (CTC) version 2.0) proteinuria, Grade 0 hematuria, and no abnormal sediment.

   Grade 0 creatinine.

   Patients must have serum creatinine within normal limits.

   Any abnormalities in the sediment or the presence of hematuria without a likely underlying cause should prompt the investigator to consider an evaluation by a nephrologist for evidence of underlying renal pathology. Patients may be eligible if the underlying cause of the abnormality is determined to be non-renal.
2. Hepatic function: Bilirubin less than 1.5 mg/dl,

   AST and ALT less than 2.5 times upper limit of normal.
3. Patients must test negative for HIV, Hepatitis B and C.

   Patients must not have other active malignancies within the past 2 years (with the exception of non-melanoma skin cancers or carcinoma in situ of the bladder) or life threatening illnesses.

   Patients must be willing to travel to the NIH for follow-up visits.

   Patients must be greater than or equal to 18 years of age.

   All patients who have received prior vaccination with vaccinia virus (for smallpox immunization) must not have a history of allergy or untoward reaction to the vaccine. Since vaccinia immunoglobulin (VIG) is available from the CDC, prior vaccinia vaccination as a safety precaution is no longer required.

   Patients must understand and sign informed consent that explains the neoplastic nature of their disease, the procedures to be followed, the experimental nature of the treatment, alternative treatments, potential risks and toxicities, and the voluntary nature of participation.

   Patients have not received the following chemotherapeutic agents for cancer within 3 years of enrolling on study: docetaxel, paclitaxel, doxorubicin, cisplatinum, carboplatinum, mitoxantrone, estramustine, cyclophosphamide, irinotecan, topotecan.

   Patients have not received prior PSA vaccine therapy.

   All patients will tested for HLA-A2. Patients must be HLA-A2+. This test may be drawn by the patient's referring physician at the time of referral (see Appendix C, HLA-typing consent). This consent will be mailed to the patient and discussed with patient. The signed consent will be signed with a witness, then mailed to the assigned research nurse at the National Institutes of Health (NIH) Clinical Center. These patients must have measurable disease on computed tomography (CT), magnetic resonance imaging (MRI), or bone scan.

   The effects of the study agents used in this protocol on the developing human fetus are unknown. For this reason men must agree to use adequate contraception prior to study entry and for the duration of study participation.

   EXCLUSION CRITERIA:

   Prior splenectomy.

   Concurrent steroid use, except topical steroids or inhaled steroid use.

   The recombinant vaccinia vaccine should not be administered if the following apply to either recipients or, for at least 3 weeks after vaccination, their close household contacts:

   persons with active or a history of eczema or other eczematoid skin disorders; those with other acute, chronic or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne or other open rashes or wounds) until condition resolves; pregnant or nursing women; children under 5 years of age; and immunodeficient or immunosuppressed persons (by disease or therapy), including HIV infection.

   Close household contacts are those who share housing or have close physical contact.

   Patients with known allergy to eggs.

   Other serious intercurrent illness.

   Patients with brain metastases.

   Patients with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment) or New York Heart Association class II-IV congestive heart failure.

   Patients on antiandrogen therapy must undergo antiandrogen withdrawal for at least 4 weeks and still show evidence of a rising PSA.

   Following treatment with bicalutamide, patients must undergo withdrawal for at least 6 weeks and still show evidence of a rising PSA.

   Prior treatments with vaccine expressing PSA are NOT eligible.

   Patients with significant autoimmune disease that is active or potentially life threatening if activated.

   Patients with clinically significant cardiomyopathy requiring treatment should be excluded from protocol eligibility at this time.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-05-22 (Actual); Primary Completion 2006-03-07 (Actual); Study Completion 2009-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Correale P, Walmsley K, Nieroda C, Zaremba S, Zhu M, Schlom J, Tsang KY. In vitro generation of human cytotoxic T lymphocytes specific for peptides derived from prostate-specific antigen. J Natl Cancer Inst. 1997 Feb 19;89(4):293-300. doi: 10.1093/jnci/89.4.293. PMID 9048833
- [Background] Vergati M, Cereda V, Madan RA, Gulley JL, Huen NY, Rogers CJ, Hance KW, Arlen PM, Schlom J, Tsang KY. Analysis of circulating regulatory T cells in patients with metastatic prostate cancer pre- versus post-vaccination. Cancer Immunol Immunother. 2011 Feb;60(2):197-206. doi: 10.1007/s00262-010-0927-9. Epub 2010 Oct 26. PMID 20976449
- [Background] Yokokawa J, Cereda V, Remondo C, Gulley JL, Arlen PM, Schlom J, Tsang KY. Enhanced functionality of CD4+CD25(high)FoxP3+ regulatory T cells in the peripheral blood of patients with prostate cancer. Clin Cancer Res. 2008 Feb 15;14(4):1032-40. doi: 10.1158/1078-0432.CCR-07-2056. PMID 18281535
- [Background] Gulley JL, Arlen PM, Madan RA, Tsang KY, Pazdur MP, Skarupa L, Jones JL, Poole DJ, Higgins JP, Hodge JW, Cereda V, Vergati M, Steinberg SM, Halabi S, Jones E, Chen C, Parnes H, Wright JJ, Dahut WL, Schlom J. Immunologic and prognostic factors associated with overall survival employing a poxviral-based PSA vaccine in metastatic castrate-resistant prostate cancer. Cancer Immunol Immunother. 2010 May;59(5):663-74. doi: 10.1007/s00262-009-0782-8. Epub 2009 Nov 5. PMID 19890632
- [Background] Stein WD, Gulley JL, Schlom J, Madan RA, Dahut W, Figg WD, Ning YM, Arlen PM, Price D, Bates SE, Fojo T. Tumor regression and growth rates determined in five intramural NCI prostate cancer trials: the growth rate constant as an indicator of therapeutic efficacy. Clin Cancer Res. 2011 Feb 15;17(4):907-17. doi: 10.1158/1078-0432.CCR-10-1762. Epub 2010 Nov 24. PMID 21106727
- [Background] Smith HA, Maricque BB, Eberhardt J, Petersen B, Gulley JL, Schlom J, McNeel DG. IgG responses to tissue-associated antigens as biomarkers of immunological treatment efficacy. J Biomed Biotechnol. 2011;2011:454861. doi: 10.1155/2011/454861. Epub 2010 Dec 19. PMID 21197272
- [Background] Kim JW, Madan RA, Gulley JL. Initial PSA oscillations precede prolonged stable disease in a patient treated with a therapeutic cancer vaccine. Clin Genitourin Cancer. 2012 Mar;10(1):43-6. doi: 10.1016/j.clgc.2011.09.003. Epub 2011 Oct 21. No abstract available. PMID 22019260
- [Result] Arlen PM, Skarupa L, Pazdur M, Seetharam M, Tsang KY, Grosenbach DW, Feldman J, Poole DJ, Litzinger M, Steinberg SM, Jones E, Chen C, Marte J, Parnes H, Wright J, Dahut W, Schlom J, Gulley JL. Clinical safety of a viral vector based prostate cancer vaccine strategy. J Urol. 2007 Oct;178(4 Pt 1):1515-20. doi: 10.1016/j.juro.2007.05.117. Epub 2007 Aug 16. PMID 17707059
- [Derived] Huang J, Jochems C, Talaie T, Anderson A, Jales A, Tsang KY, Madan RA, Gulley JL, Schlom J. Elevated serum soluble CD40 ligand in cancer patients may play an immunosuppressive role. Blood. 2012 Oct 11;120(15):3030-8. doi: 10.1182/blood-2012-05-427799. Epub 2012 Aug 28. PMID 22932804
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: Drug Information Portal — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 32 patients were accrued to the phase II portion of the study
Groups:
- no GM: Vaccine subcutaneously with no GM
- Rec-hGM: Vaccine subcutaneously with Rec-hGM sucutaneously (daily x 4/vaccine)
- rF-GM (10^7pfu): Vaccine subcutaneously with rF-GM (10^7pfu) subcutaneously x1
- rF-GM (10^8): Vaccine subcutaneously with rF-GM (10^8) subcutaneously x1
Period: Overall Study
Arm/Group | no GM | Rec-hGM | rF-GM (10^7pfu) | rF-GM (10^8)
Started | 8 (32 participants are reported for the phase II portion.) | 9 | 7 | 8
Completed | 8 | 9 | 7 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prostate Cancer Patients: Progressive Metastatic Castration Resistant Prostate Cancer
Arm/Group | Prostate Cancer Patients
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 32
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Immune Response
Description: Immune response is defined as an enhanced PSA specific T-cell immune response greater than or equal to twofold post-vaccination. Peripheral blood mononuclear cells (PBMCs) were collected by apheresis prior to treatment with vaccination and after approximately three months of therapy.
Time Frame: 48 months
Measure: Count of Participants; unit: Participants
Groups:
- rF-GM (10^7pfu),: Vaccine subcutaneously with rF-GM (10^7pfu) subcutaneously x1
Arm/Group | No GM | Rec-hGM | rF-GM (10^7pfu), | rF-GM (10^8)
Number analyzed (Participants) | 8 | 6 | 7 | 8
Participants | 2 | 4 | 4 | 3

2. Secondary Outcome: Percent of Participants With a Decrease (i.e. Greater Than or Equal to 30%) in PSA Levels
Description: PSA level at the time treatment is initiated compared to the PSA level at Day 85 and monthly thereafter while the patient continues on trial)
Time Frame: 53 months
Population: PSA was taken at multiple time points and proportion of patients (pts) who had a decrease in PSA of at least 30% was reported. This is standard reporting procedures for tumor markers (proportion of patients with a response);similar to RECIST reporting where there may be multiple scans obtained but one reports the proportion of pts with a response
Measure: Number; unit: Percentage of participants
Groups:
- Phase 2: Phase 2 patients are randomized between 4 arms:e.g. No GM, Rec-hGM, rF-GM (10^7pfu), rF-GM (10^8) with efficacy and immunological response as a primary endpoint.
Arm/Group | Phase 2
Number analyzed (Participants) | 32
Percentage of participants | 15.6

3. Secondary Outcome: Number of Participants With an Objective Response
Description: Objective response is determined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria defined as: measurable disease (at least one measurable lesion), measurable lesions (lesions that can be accurately measured in at least one dimension with longest diameter >/= 20 mm using conventional techniques or >/= 10 mm with spiral CT scan. Non-measurable lesions (all other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan), i.e. bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusion...
Time Frame: 53 months
Population: All 12 participants with measurable disease were evaluated.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2: Phase 2 patients are randomized between 4 arms: e.g. No GM, Rec-hGM, rF-GM (10^7pfu), rF-GM (10^8) with efficacy and immunological response as a primary endpoint.
Arm/Group | Phase 2
Number analyzed (Participants) | 12
Participants | 0

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the date of on-study to the date of death from any cause or last follow-up.
Time Frame: 50 months
Measure: Median (Full Range); unit: Months
Groups:
- Phase 2: Phase 2 patients are randomized between 4 arms: e.g. No GM, Rec-hGM, rF-GM (10^7pfu), rF-GM (10^8)with efficacy and immunological response as a primary endpoint.
Arm/Group | Phase 2
Number analyzed (Participants) | 32
Months | 26.6 [6 to 50]

5. Secondary Outcome: The Number of Participants With Adverse Events
Description: Here are the total number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 77.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2
Number analyzed (Participants) | 32
Participants | 32

ADVERSE EVENTS:
Time Frame: 77.5 months
Arm/Group | no GM | Rec-hGM | rF-GM (10^7pfu) | rF-GM (10^8)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 3/9 | 2/7 | 3/8
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 7/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | no GM (N=8) | Rec-hGM (N=9) | rF-GM (10^7pfu) (N=7) | rF-GM (10^8) (N=8)
Supraventricular arrhythmias (supraventricular tachycardia (SVT)/atrial fibrillation/flutter) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constitutional Symptoms-Other (Specify_) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Death 9 months post last vaccine 4/5/04
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mood alteration-depression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | no GM (N=8) | Rec-hGM (N=9) | rF-GM (10^7pfu) (N=7) | rF-GM (10^8) (N=8)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 4 (5) | 0 (0) | 3 (5) | 1 (2)
Creatinine (Renal and urinary disorders) | 3 (7) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (5) | 1 (1) | 1 (1)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 4 (6) | 4 (9) | 2 (5) | 3 (3)
Bruising (in absence of grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 7 (30) | 8 (20) | 6 (40) | 7 (21)
Rash/desquamation (Social circumstances) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (4)
Hypoalbuminemia (Hepatobiliary disorders) | 4 (5) | 4 (6) | 5 (17) | 7 (9)
SGPT (ALT) (serum glutamic pyruvic transaminase) (alanine aminotransferase) (Hepatobiliary disorders) | 3 (3) | 0 (0) | 3 (5) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (14) | 7 (11) | 6 (13) | 3 (6)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 1 (2) | 1 (2) | 1 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (6) | 3 (5) | 3 (3) | 2 (2)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (aspartate aminotransferase) (Hepatobiliary disorders) | 5 (5) | 3 (4) | 5 (9) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (3) | 4 (5) | 2 (3)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 4 (10) | 4 (5) | 5 (12) | 3 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain or cramping (Reproductive system and breast disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 2 (3) | 1 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inner ear/hearing (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytes (total white blood cell (WBC)) (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasovagal episode (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema (Cardiac disorders) | 2 (3) | 0 (0) | 2 (2) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prothrombin time (PT) (Congenital, familial and genetic disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Rigors, chills (General disorders) | 1 (1) | 2 (5) | 2 (4) | 0 (0)
Sweating (diaphoresis) (General disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (3)
Weight loss (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Wound-non-infectious (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dysphagia, esophagitis, odonphagia (painful swallowing) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Mouth dryness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (in the absence of vaginal bleeding) (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase (Hepatobiliary disorders) | 3 (3) | 3 (5) | 4 (5) | 3 (4)
Bilirubin (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infection without neutropenia (Infections and infestations) | 2 (6) | 5 (5) | 2 (4) | 0 (0)
Bicarbonate (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hypermagnesemia (Musculoskeletal and connective tissue disorders) | 1 (4) | 3 (3) | 2 (3) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 2 (4) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness/lightheadedness (Nervous system disorders) | 2 (4) | 2 (4) | 1 (2) | 2 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 2 (2) | 1 (1)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (fainting) (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia/heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sense of smell (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mood alteration/depression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (non-cardiac and non-pleuritic) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Earache (otalgia) (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Reproductive system and breast disorders) | 0 (0) | 3 (4) | 1 (3) | 0 (0)
Pain-Other (Specify_) (General disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0) — 1. Pain rt-hip 2. pain in testicles 3. groin pain 4. pain: tongue "raw" 5. Back pain
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis/embolism (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Nervous system disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Mood alteration-anxiety, agitation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy-sensory (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syndromes-Other (Specify-flu like syndrome) (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dermatology/Skin-Other (Specify_) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — 1. At vaccine site 3 cm firmness 2. derm: induration "knot" 3. small growth on anal
Epistaxis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 4 (7) | 4 (5) | 4 (5) | 7 (12)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC <1.0x10e9/L) (General disorders) | 1 (1) | 3 (3) | 1 (2) | 2 (5)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (3)
Ventricular arrhythmia (PVCs/bigeminy/trigeminy/ventricular tachycardia) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Diarrhea patients with a colostomy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection without neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysuria (painful urination) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bicarbonate (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No